CLINICAL TRIAL: NCT01368835
Title: Evaluation of the Ulthera™ System For Obtaining Lift and Tightening of the Cheek Tissue and Improvement in Jawline Definition and Submental Skin Laxity
Brief Title: Evaluation of the Ulthera™ System for Obtaining Lift and Tightening of the Cheek Tissue
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ulthera, Inc (Industry)
Collaborators: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Organization: Merz North America, Inc. (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: ULT-106
Record Dates: First submitted 2011-06-06; First posted 2011-06-08 (Estimated); Results first posted 2013-08-15 (Estimated); Last update posted 2017-12-13 (Actual); Status verified 2014-01

CONDITIONS: Mild to Moderate Skin Laxity on Cheek; Mild to Moderate Skin Laxity on Upper Neck; Mild to Moderate Subcutaneous Fat on Cheek; Mild to Moderate Subcutaneous Fat on Upper Neck

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Ulthera treatment (Experimental)
  Interventions: Device: Ulthera treatment

INTERVENTIONS:
Device: Ulthera treatment — treatment of cheeks and upper neck area of face

SUMMARY:
The clinical trial evaluates the clinical outcomes associated with the non-invasive treatment to obtain lift and tightening of the cheek tissue and improve jawline definition and submental skin laxity utilizing the Ulthera™ System which delivers ultrasound energy in a focused manner below the surface of the skin

DETAILED DESCRIPTION:
The primary objective of this study is to demonstrate the effectiveness of the Ulthera™ System for the non-invasive dermatological treatment to obtain lift and tighten the cheek tissue.

The secondary objective of this study is to demonstrate the effectiveness of the Ulthera™ System for the non-invasive dermatological treatment for improvement in jawline definition and submental skin laxity at 3 and 6 months compared to baseline based on the consensus of the three masked reviewers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged 35 to 60 years
* Subject in good health
* Desire lift and tightening of cheek tissue, improvement of jawline definition or submental skin laxity

Exclusion Criteria:

* Pregnant or lactating
* Has an active systemic or local skin disease that may alter wound healing
* Severe solar elastosis
* Excessive subcutaneous fat on the cheeks
* Excessive skin laxity on the lower face and neck
* Has significant scarring in areas to be treated
* Has significant open facial wounds or lesions
* Has severe or cystic acne on the face

Ages: 35 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 103 (Actual)
Dates: Start 2010-07; Primary Completion 2010-12 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey M. Kenkel, MD, Principal Investigator — University of Texas Southwestern Medical Center

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment from June 30, 2010 to August 31, 2010.
Pre-assignment Details: Male or Female, aged 30 to 60 years. Desire to lift and tighten cheek tissue, improve jawline definition and/or submental skin laxity.
Groups:
- Ulthera Treatment: Subjects will receive one dual-depth focused ultrasound treatment to their lower face and submental regions.
Period: Overall Study
Arm/Group | Ulthera Treatment
Started | 103 (103 Subjects Enrolled)
Completed | 70
Not Completed | 33
Not completed — Inclusion criteria/photography quality | 22
Not completed — Lost to Follow-up | 11

BASELINE CHARACTERISTICS:
Population: N=33 Excluded from analysis: N=22 excluded for inclusion criteria/photo lighting/positional/makeup issues and N=11 lost to follow-up.
Groups:
- Ulthera Treatment: Treatment to the lower face and submental region.
Arm/Group | Ulthera Treatment
Number analyzed (Participants) | 70
Age, Continuous [Mean (Full Range); unit: years] — Average patient age
  years | 49.5 [35 to 58]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57
  Male | 13
Region of Enrollment [Number; unit: participants]
  United States | 70
Fitzpatrick Skin Type [Number; unit: # of Participants] — Skin Type I = White; very fair, red or blonde hair blue eyes; freckles; Always burns, never tans
  Skin Type II = White, fair, red or blond hair; blue, hazel or green eyes; Usually burns, tans with difficulty
  Skin Type III = Cream white; fair with any eye or hair color (common); Sometimes mild burn, gradually tans
  Skin Type IV = Brown; typical Mediterranean Caucasian skin; Rarely burns, tans with ease
  Skin Type V = Dark Brown; mid-eastern skin types; Very rarely burns, tans easily
  Skin Type VI = Black; Never burns, tans very easily
  # of Participants
    Skin Type I | 9
    Skin Type II | 46
    Skin Type III | 12
    Skin Type IV | 2
    Skin Type V | 1

OUTCOME MEASURES:

1. Primary Outcome: Change in Overall Lifting and Tightening of Treated Tissue on the Lower Face and Submental Regions.
Description: The percentage of participants assessed to have improvement in skin laxity, i.e., lifted and tightened skin in the areas treated with the Ulthera System, as determined by three masked assessors comparing pre-treatment and 90-days post-treatment photos from 70 subjects who returned for their 90-day follow-up visit.
Time Frame: 90D
Population: The number of participants who received an Ulthera treatment and for whom pre-treatment and 90-day post-treatment photos were available, i.e., evaluable participants, for a masked assessment.
Measure: Number; unit: percentage of participants improved
Groups:
- Ulthera Treatment: Subjects who received one focused ultrasound treatment to the lower face and submental regions using the Ultera System.
Arm/Group | Ulthera Treatment
Number analyzed (Participants) | 70
percentage of participants improved | 68.60

2. Secondary Outcome: Change in Submental and Neck Skin Laxity by Quantitative Analysis
Description: The percentage of participants assessed as having an improvement in tissue lift, i.e., >20mm2 in submental and neck skin laxity, at 90 Days post-treatment compared to baseline based on quantitative analysis.
Time Frame: 90D
Population: The number of participants who received an Ulthera treatment and for whom pre-treatment and 90-day post-treatment photos were available, i.e., evaluable participants.
Measure: Number; unit: percentage of participants improved
Arm/Group | Ulthera Treatment
Number analyzed (Participants) | 70
percentage of participants improved | 72.9

3. Secondary Outcome: Patient Satisfaction Questionnaire
Description: Subjects indicated whether they saw improvement, i.e., providing a Yes/No response, in face and neck characteristics at three months (D90) post Ulthera treatment. Pre-treatment and Day 90 post-treatment photographs were available for viewing during the assessment. Subjects also had a mirror in hand for real time assessment. Subjects' Yes/No responses were tabulated.
Time Frame: 90D
Population: The number of participants who received an Ulthera treatment and for whom pre-treatment and 90-day post-treatment photos were available.
Measure: Number; unit: percentage of participants improved
Arm/Group | Ulthera Treatment
Number analyzed (Participants) | 70
percentage of participants improved | 67

4. Other Pre Specified Outcome: Subject Assessment of Pain
Description: Subject assessment of pain using a validated Numeric Rating Scale (NRS), 0-10, where 0 = no pain and 10=worse pain possible. Subjects' sensory responses to the treatment exposures were recorded using the NRS for each anatomical region.
Time Frame: During Ulthera study treatment
Population: Evaluable subjects, i.e., n=70, who received an Ulthera treatment and for whom an NRS was completed.
Measure: Mean (Full Range); unit: Average NRS score
Arm/Group | Ulthera Treatment
Number analyzed (Participants) | 70
Average NRS score | 6.13 [1 to 10]

ADVERSE EVENTS:
Time Frame: Baseline, Treatment, D90, D180
Description: Device and/or procedure related adverse events
Arm/Group | Ulthera Treatment
Serious Adverse Events (participants affected / at risk) | 0/103
Other Adverse Events (participants affected / at risk) | 0/103

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less